CLINICAL TRIAL: NCT01699581
Title: Assessment of Impact Nutritional Program During Autologous Stem Cell Transplant
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Research cancelled following interim analysis
Sponsor: Greg Monohan (Other)
Responsible Party: Sponsor-Investigator, Greg Monohan, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-HEM-03-MCC
Record Dates: First submitted 2012-09-27; First posted 2012-10-03 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Hodgkin's Lymphoma; Multiple Myeloma; Non-Hodgkin's Lymphoma
Keywords: Hodgkin's Lymphoma; Multiple Myeloma; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Multiple Myeloma; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nestle Impact Advanced Recovery (Experimental): Nestle Impact Advanced Recovery
  1 dose of Nestle Impact Advanced Recovery orally three times a day
  Interventions: Dietary Supplement: Nestle Impact Advanced Recovery

INTERVENTIONS:
Dietary Supplement: Nestle Impact Advanced Recovery — dose of Nestle Impact Advanced Recovery orally three times a day beginning on the morning following stem cell transplant and continued until the day of hospital discharge.

SUMMARY:
Nestle Impact has shown efficacy in multiple surgical trials in relation to improving hospital length of stay and infection rate. 1 dose of Nestle Impact Advanced Recovery will be taken orally three times a day beginning on the morning following stem cell transplant and will continue until the day of hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving an autologous stem cell transplant using the preparative regimens of BEAM (Carmustine, Etoposide, Cytarabine, Melphalan), Melphalan 140mg/m2, or Melphalan 200mg/m2
* Any prior diet or supplement will be allowed.
* Age >18 years.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Nestle Impact including fish oil.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-09; Primary Completion 2014-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Hospital length of stay | Particpants will be followed for 14 days, the average length of time from stem cell infusion until dischcarge
Days to engraftment | Particpants will be followed for 14 days, the average length of time from stem cell infusion until dischcarge

CONTACTS AND LOCATIONS:
Overall Officials: Greg Monohan, MD, Principal Investigator — Lucille P. Markey Cancer Center at University of Kentucky
Locations (1):
- University of Kentucky, Markey Cancer Center, Lexington, Kentucky, United States